CLINICAL TRIAL: NCT00361374
Title: Omega-3 Fatty Acids for Treatment of Major Depression: Differential Effects of EPA and DHA, and Associated Biochemical and Immune Parameters
Brief Title: Safety and Effectiveness of Omega 3-Fatty Acids, EPA Versus DHA, for the Treatment of Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Cedars-Sinai Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Mischoulon, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005P002337; 5R01MH074085 (NIH)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Omega-3; Boston
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Eicosapentaenoic Acid; Fatty Acids, Omega-3; Docosahexaenoic Acids; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EPA (Experimental): Eicosapentaenoic acid (EPA) Omega-3, 1g/day
  Interventions: Dietary Supplement: eicosapentaenoic acid
- DHA (Experimental): Docosahexaenoic acid (DHA) Omega-3, 1g/day
  Interventions: Dietary Supplement: docosahexaenoic acid
- Placebo (Placebo Comparator): Placebo capsule (980mg soybean oil)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: eicosapentaenoic acid — 1 gram/day
  Other Names: EPA, Omega-3 Fatty Acid, ProEPAXtra
  Arms: EPA
Dietary Supplement: docosahexaenoic acid — 1 gram/day
  Other Names: DHA, Omega-3 Fatty Acid, ProDHA
  Arms: DHA
Drug: Placebo — 980 milligram/day
  Other Names: Placebo, Soybean oil
  Arms: Placebo

SUMMARY:
This study examines the difference in the effectiveness of two natural compounds, eicosapentanoic (EPA) and docosahexanoic (DHA)omega-3 fatty acids, in treating major depressive disorder. Both types of omega-3 fatty acids are commonly found in fish oils. It is believed that a deficiency in these omega-3 fatty acids may lead to the development of major depression.

DETAILED DESCRIPTION:
The study lasts for eight weeks and involves four visits after the screen and baseline visits (biweekly). Participants will be randomized, or chosen by chance, to enter into one of three groups. People in the first group will take 1 g/day or EPA omega-3 fatty acid, those in the second group will take 1 g/day of DHA omega-3 fatty acid, and those in the third group will take a placebo. This study is double-blind, which means that neither the participant, nor the doctor, nor the research staff will know which group each person is in. At the end of the study the participant will be offered three months of follow-up care at the Depression Clinical and Research Program.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-80 years old.
* Must meet criteria for current Major Depressive Disorder.

Exclusion Criteria:

* Serious or unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease
* History of seizure disorder.
* Substance use disorders, including alcohol, active within the last six months (past history is OK).
* History of multiple adverse drug reactions or allergy to the study drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2006-07; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mischoulon, MD, PhD, Principal Investigator — Depression Clinical and Research Program, Massachusetts General Hospital
Locations (1):
- Depression Clinical Research Program, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851
- See also: The Depression Clinical and Research Program at Massachusetts General Hospital — http://www.massgeneral.org/depression

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 196 adults with MDD were recruited from 05/18/06 to 06/30/11 at Massachusetts General Hospital and Cedars-Sinai Medical Center.
Groups:
- Eicosapentaenoic Acid (EPA): Eicosapentaenoic acid (EPA) Omega-3, 1g/day
  eicosapentaenoic acid: 1 gram/day
- Docosahexaenoic Acid (DHA): Docosahexaenoic acid (DHA) Omega-3, 1g/day
  docosahexaenoic acid: 1 gram/day
Period: Overall Study
Arm/Group | Eicosapentaenoic Acid (EPA) | Docosahexaenoic Acid (DHA) | Placebo
Started | 66 | 65 | 65
Completed | 51 | 50 | 53
Not Completed | 15 | 15 | 12

BASELINE CHARACTERISTICS:
Population: We randomized 196 of 389 screened patients. Nineteen subjects dropped out before completing at least one post-baseline visit, leaving 177 evaluable subjects for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eicosapentaenoic Acid (EPA) | Docosahexaenoic Acid (DHA) | Placebo | Total
Number analyzed (Participants) | 60 | 58 | 59 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12.5) | 46.2 (11.8) | 45.0 (12.1) | 45.8 (12.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 50 | 54 | 157
  >=65 years | 7 | 8 | 5 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 35 | 105
  Male | 22 | 26 | 24 | 72
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 59 | 177

OUTCOME MEASURES:

1. Primary Outcome: Score on a Depression Severity Rating Scale Over Eight Weeks
Description: Change in score on 17-item Hamilton D depression severity rating scale over 8 weeks of treatment. Scores were obtained every 2 weeks for 8 weeks. The total sum score of the 17 items is used to assess depressive severity. Possible total scores range from 0-52, with a higher score indicating greater depressive severity. Scores of 7 or less are indicative of full remission (i.e. no depression). Scores of 8-15 indicate mild depression; scores of 16-25 indicate moderate depression; scores of 25 or greater indicate severe depression. Mixed model repeated measures analysis (MMRM) was used to examine treatment group effect on changes from baseline to week 8 in Hamilton D scores. Models included subjects as a random effect, and treatment group and study week as fixed effects. An auto-regressive covariance structure was used because it provided the best fit to the data. Site and baseline score were included as covariates in all models.
Time Frame: 8 weeks
Population: We randomized 196 of 389 screened patients. Nineteen subjects dropped out before completing at least one post-baseline visit, leaving 177 evaluable subjects
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Eicosapentaenoic Acid (EPA) | Docosahexaenoic Acid (DHA) | Placebo
Number analyzed (Participants) | 60 | 58 | 59
units on a scale | -10.34 (0.62) | -9.26 (0.62) | -9.49 (0.61)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 8 weeks of the study period.
Arm/Group | Eicosapentaenoic Acid (EPA) | Docosahexaenoic Acid (DHA) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 39/60 | 40/58 | 43/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eicosapentaenoic Acid (EPA) (N=60) | Docosahexaenoic Acid (DHA) (N=58) | Placebo (N=59)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 8 (8) | 11 (11)
Constipation (Gastrointestinal disorders) | 8 (8) | 8 (8) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 7 (7) | 4 (4)
Nausea or vomiting (Gastrointestinal disorders) | 7 (7) | 8 (8) | 5 (5)
Palpitations (Cardiac disorders) | 8 (8) | 7 (7) | 2 (2)
Dizziness on standing (Cardiac disorders) | 5 (5) | 7 (7) | 4 (4)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Increased perspiration (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 4 (4)
Itching (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7) | 8 (8)
Headache (Nervous system disorders) | 8 (8) | 12 (12) | 12 (12)
Tremors (Nervous system disorders) | 1 (1) | 5 (5) | 0 (0)
Poor coordination (Nervous system disorders) | 2 (2) | 6 (6) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 7 (7) | 4 (4)
Blurred vision (Eye disorders) | 5 (5) | 5 (5) | 7 (7)
Ringing in ears (Ear and labyrinth disorders) | 4 (4) | 2 (2) | 2 (2)
Difficulty urinating (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Painful urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Frequent urination (Renal and urinary disorders) | 9 (9) | 5 (5) | 3 (3)
Menstrual irregularity (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 3 (3)
Difficulty sleeping (Psychiatric disorders) | 18 (18) | 11 (11) | 12 (12)
Sleeping too much (Psychiatric disorders) | 4 (4) | 7 (7) | 6 (6)
Loss of sexual desire (Psychiatric disorders) | 7 (7) | 9 (9) | 12 (12)
Trouble achieving orgasm (Psychiatric disorders) | 6 (6) | 3 (3) | 2 (2)
Trouble with erections (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 10 (10) | 14 (14) | 14 (14)
Poor concentration (Psychiatric disorders) | 13 (13) | 12 (12) | 14 (14)
General malaise (Psychiatric disorders) | 5 (5) | 7 (7) | 12 (12)
Restlessness (Psychiatric disorders) | 4 (4) | 8 (8) | 12 (12)
Fatigue (Psychiatric disorders) | 14 (14) | 13 (13) | 9 (9)
Decreased energy (Psychiatric disorders) | 16 (16) | 12 (12) | 13 (13)

LIMITATIONS AND CAVEATS:
The study was underpowered due to lower than expected recruitment. The high placebo response rate may have impeded signal detection. The n-3 preparations were not pure, but "enriched" for one n-3 or the other, and contained other FAs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No